CLINICAL TRIAL: NCT04839133
Title: Feasibility of Robotic Assisted Exercise Training in Patients With Advanced Heart Failure or Advanced Pulmonary Diseases
Brief Title: Robotic-assisted Exercise Training in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Heart Institute (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MyoSuit Feasibility Trial
Record Dates: First submitted 2021-03-29; First posted 2021-04-09 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure, Systolic; Pulmonary Disease
Keywords: Exercise training; Robotic training; Exosuit training
MeSH Terms: conditions — Heart Failure, Systolic; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility study group (Other)
  Interventions: Device: MyoSuitFeasibility

INTERVENTIONS:
Device: MyoSuitFeasibility — Participants will absolve feasibility tests with and without wearing a MyoSuit.

SUMMARY:
Background:

Regular physical activity is an evidence-based adjuvant therapy of chronic heart failure or chronic lung diseases. Structured exercise training is safe, increases exercise capacity and quality of life, relieves symptoms and reduces hospitalization rates. Even a trend towards reduction of mortality has been identified. However, dyspnea and fatigue, typical symptoms of heart or lung failure, force patients to physical inactivity which fatally aggravates deconditioning and exercise intolerance, leading to an increased risk of hospitalization and a loss of independence and quality of life. To break through this vicious circle physical activity must be restored, since exercise intolerance can be successfully improved by physical training.

Purpose:

This study will address the challenging task of remobilizing patients with advanced chronic lung or heart failure in a functional New York Heart Association class III-IV by using an externally physically-supported exosuit movement therapy. This soft, wearable robot (fig. 1) assists mobilization according to individual needs by activating neuromuscular feedback systems, promoting physical activity and preventing early physical exhaustion. The investigators hypotheses that an exosuit-supported training increases exercise capacity and quality of life in a greater degree than non-supported training.

Methods:

The study will consist of two parts investigating i) the feasibility, tolerance and safety (n= 30) and ii) the efficacy of an exosuit device-supported training (n=30). In i) patients will perform a walking test and a set of everyday life skills or participate in a standardized rehabilitation sports program. In ii) patients will be randomized in a 2:1 ratio for an exosuit-supported or non-supported exercise training protocol, training 3 units per week for 8 weeks. Assessment of outcome will be performed by various functional, mobility and endurance tests, questionnaires and clinical parameters. Furthermore, the transfer of regained motor and balance skills to everyday life will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* >17 years old
* written informed consent
* chronic end-stage systolic heart failure without ventricular assist device, LVEF ≤ 45% OR chronic advanced pulmonary diseases
* clinically stable for at least 6 weeks
* ability to mobilize into standing and walking of at least 10 meters with or without rollator
* ability to get up from a chair without rotating the upper body >45° sagittally

Exclusion Criteria:

* addictions or other illnesses that impact the ability to understand the nature, scope and consequences of the trial
* lack of knowledge of German to fully understand study information
* pregnancy, pre-menopausal women
* contraindications of cardiopulmonary exercising
* BMI > 35 kg/m², waist size > 135 cm.
* Height <150 cm, >195 cm
* Weight<45 kg, >110 kg
* Functional Reach Test <15,24 cm
* Flexion contracture in the knee/hip joint >10°
* Chronic colonization or active infection with multi-resistant pathogens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Falls - Safety of the MyoSuit | 1 hour
  Patients with advanced heart or pulmonary failure will perform 6-minute walking tests and activities of daily life both with and without wearing a MyoSuit. Outcome is measured by documenting number of falls.
Incidence of Treatment-Emergent Adverse Events - Safety of the MyoSuit | 1 hour
  Patients with advanced heart or pulmonary failure will perform 6-minute walking tests and activities of daily life both with and without wearing a MyoSuit. Outcome is measured by documenting adverse events.
Exercise can be performed when wearing a MyoSuit - Feasibility and Tolerability of walking test, activities of daily life, rehabilitation exercise group. | 1 hour
  Patients with advanced heart or pulmonary failure will perform a 6 minute walking test, activities of daily life and a cardiac rehabilitation exercise unit. Outcome is measured dichotomously (yes/no) according to its feasibility.
Necessity of assistance in exercising when wearing a MyoSuit - Feasibility and Tolerability | 1 hour
  Patients with advanced heart or pulmonary failure will perform a 6 minute walking test, activities of daily lif and a cardiac rehabilitation exercise unit. Outcome is measured according to a scale of assistance needed (1=no assistance, 2=little assistance, 3=much assistance, 4=not possible). 1 is minimum, 4 is maximum. The higher the score, the worse the outcome.
MyoSuit assistance leads to changes in walking distance in patients with advanced heart or pulmonary failure assessed by 6-minute walking test. | 30 minutes
  Change of 6minute walk distance in meters will be assessed with and without MyoSuit in every participant.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - German Heart Center, Berlin
  - German Heart Institute, Berlin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Just IA, Fries D, Loewe S, Falk V, Cesarovic N, Edelmann F, Feuerstein A, Haufe FL, Xiloyannis M, Riener R, Schoenrath F. Movement therapy in advanced heart failure assisted by a lightweight wearable robot: a feasibility pilot study. ESC Heart Fail. 2022 Jun;9(3):1643-1650. doi: 10.1002/ehf2.13903. Epub 2022 Mar 23. PMID 35320878